CLINICAL TRIAL: NCT01498133
Title: Does Skin-to-skin Contact Promote Bacterial Decolonization in Preterm Infants in Neonatal Intensive Care Unit? A Randomized, Single-blinded Controlled Trial
Brief Title: Skin-to-skin Contact to Promote Bacterial Decolonization in Preterm Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Maranhão (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fernando Lamy Filho, Principal Investigator, Universidade Federal do Maranhão
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2011-11-21; First posted 2011-12-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: PREMATURITY
Keywords: Skin-to-skin contact; Decolonization; MRSA
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- skin-to-skin contact (Experimental): Newborns in the study group had skin-to-skin contact with their mothers in the NICU, twice a day (morning and evening) for 60 minutes, for seven days (including weekends).
  Interventions: Procedure: skin-to skin contact
- control group (No Intervention): The control group (n = 49) received routine care without skin-to-skin contact.

INTERVENTIONS:
Procedure: skin-to skin contact — Skin-to-skin contact consisted of placing the infant slightly worn (only diapers) in prone decubitus, upright against the mother's breast. The infant was restrained in position by a track that involved him with his/her mother. The mother sat in a chair positioned beside the infants' bed. A team member that accompanied the intervention monitored infants' temperature, heart rate and oxygen saturation.
  Other Names: Kangaroo mother care
  Arms: skin-to-skin contact

SUMMARY:
BACKGROUND Decolonization with topical antibiotics is necessary to prevent and / or control outbreaks of multidrug-resistant bacterial infection in the NICU (Neonatal Intensive Care Unit), but can trigger bacterial resistance. The objective of this study was to determine whether skin-to-skin contact of newborns colonized with MRSA (Methicillin-Oxacillin Resistant Staphylococcus Aureus) with their mothers could be an effective alternative for biological control of bacterial colonization.

METHODS: The investigators studied 102 newborns admitted to NICU in three public hospitals in São Luís, Brazil. Inclusion criteria were birth weight from 1300 to 1800g, length of stay >4 days, newborns colonized by Staphylococcus aureus and/or Staphylococcus coagulase-negative methicillin-oxacillin resistant and mothers not colonized by these bacteria. Randomization was performed using a computer generated random numbers algorithm. Allocation to intervention and control groups was performed for each eligible newborn using a sealed opaque envelope. In the intervention group (n = 53) mother-infant skin-to-skin contact was held twice a day. The control group (n = 49) received routine care without skin-to-skin contact. There was no masking of newborn's mothers or researchers, but the individuals who carried out bacterial cultures and assessed results were kept blind to group allocation.

The primary outcome was decolonization of newborns' nostrils after 7 days of intervention. Safety was assessed by monitoring vital signs of newborns during the intervention. The secondary outcome was emergence of late onset presumed sepsis until the end of hospitalization period or 28 days of life, whatever happened first.

FUNDING: CNPq (Brazilian Research Council) and FAPEMA (Maranhão Research Foundation)

ELIGIBILITY:
Inclusion Criteria:

* singleton neonates,
* born in the three institutions of the study
* birth weight from 1300 to 1800g
* length of stay >=4 days,
* newborns colonized by Staphylococcus aureus and/or Staphylococcus coagulase-negative methicillin-oxacillin resistant and mothers not colonized by these bacterias.

Exclusion Criteria:

* infants below 1300g and over 1800g,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Decolonization of newborns' nostrils | 7 days
  The primary outcome was decolonization of newborns' nostrils after 7 days of intervention

SECONDARY OUTCOMES:
late onset presumed sepsis | The end of hospitalization period or 28 days of life, whatever happened first.
  The secondary outcome was emergence of late onset presumed sepsis until the end of hospitalization period or 28 days of life, whatever happened first.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Lamy Filho, PhD, Principal Investigator — Universidade Federal do Maranhao - Programa de Posgraduação em Saúde Coletiva
Locations (1):
- Hospital Universitario Da Universidade Federal Do Maranhao, São Luís, Maranhão, Brazil

REFERENCES:
- [Background] Morel AS, Wu F, Della-Latta P, Cronquist A, Rubenstein D, Saiman L. Nosocomial transmission of methicillin-resistant Staphylococcus aureus from a mother to her preterm quadruplet infants. Am J Infect Control. 2002 May;30(3):170-3. doi: 10.1067/mic.2002.119819. PMID 11988712
- [Background] Humphreys H. Can we do better in controlling and preventing methicillin-resistant Staphylococcus aureus (MRSA) in the intensive care unit (ICU)? Eur J Clin Microbiol Infect Dis. 2008 Jun;27(6):409-13. doi: 10.1007/s10096-008-0469-7. Epub 2008 Feb 13. PMID 18270758
- [Background] Gerber SI, Jones RC, Scott MV, Price JS, Dworkin MS, Filippell MB, Rearick T, Pur SL, McAuley JB, Lavin MA, Welbel SF, Garcia-Houchins S, Bova JL, Weber SG, Arnow PM, Englund JA, Gavin PJ, Fisher AG, Thomson RB, Vescio T, Chou T, Johnson DC, Fry MB, Molloy AH, Bardowski L, Noskin GA. Management of outbreaks of methicillin-resistant Staphylococcus aureus infection in the neonatal intensive care unit: a consensus statement. Infect Control Hosp Epidemiol. 2006 Feb;27(2):139-45. doi: 10.1086/501216. Epub 2006 Feb 8. PMID 16465630
- [Background] Uehara Y, Kikuchi K, Nakamura T, Nakama H, Agematsu K, Kawakami Y, Maruchi N, Totsuka K. Inhibition of methicillin-resistant Staphylococcus aureus colonization of oral cavities in newborns by viridans group streptococci. Clin Infect Dis. 2001 May 15;32(10):1399-407. doi: 10.1086/320147. Epub 2001 Apr 17. PMID 11317239
- [Background] Shimizu A, Shimizu K, Nakamura T. Non-pathogenic bacterial flora may inhibit colonization by methicillin-resistant Staphylococcus aureus in extremely low birth weight infants. Neonatology. 2008;93(3):158-61. doi: 10.1159/000108413. Epub 2007 Sep 18. PMID 17878742
- [Background] Kawada M, Okuzumi K, Hitomi S, Sugishita C. Transmission of Staphylococcus aureus between healthy, lactating mothers and their infants by breastfeeding. J Hum Lact. 2003 Nov;19(4):411-7. doi: 10.1177/0890334403257799. PMID 14620455
- [Background] Sakaki H, Nishioka M, Kanda K, Takahashi Y. An investigation of the risk factors for infection with methicillin-resistant Staphylococcus aureus among patients in a neonatal intensive care unit. Am J Infect Control. 2009 Sep;37(7):580-6. doi: 10.1016/j.ajic.2009.02.008. Epub 2009 Jun 17. PMID 19535174
- [Background] Goetghebeur M, Landry PA, Han D, Vicente C. Methicillin-resistant Staphylococcus aureus: A public health issue with economic consequences. Can J Infect Dis Med Microbiol. 2007 Jan;18(1):27-34. doi: 10.1155/2007/253947. PMID 18923684
- [Background] Huang YC, Chou YH, Su LH, Lien RI, Lin TY. Methicillin-resistant Staphylococcus aureus colonization and its association with infection among infants hospitalized in neonatal intensive care units. Pediatrics. 2006 Aug;118(2):469-74. doi: 10.1542/peds.2006-0254. PMID 16882797
- [Background] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics. 2002 Aug;110(2 Pt 1):285-91. doi: 10.1542/peds.110.2.285. PMID 12165580
- [Background] Moss W, Darmstadt GL, Marsh DR, Black RE, Santosham M. Research priorities for the reduction of perinatal and neonatal morbidity and mortality in developing country communities. J Perinatol. 2002 Sep;22(6):484-95. doi: 10.1038/sj.jp.7210743. PMID 12168128
- [Background] McConeghy KW, Mikolich DJ, LaPlante KL. Agents for the decolonization of methicillin-resistant Staphylococcus aureus. Pharmacotherapy. 2009 Mar;29(3):263-80. doi: 10.1592/phco.29.3.263. PMID 19249946
- [Background] Pinter DM, Mandel J, Hulten KG, Minkoff H, Tosi MF. Maternal-infant perinatal transmission of methicillin-resistant and methicillin-sensitive Staphylococcus aureus. Am J Perinatol. 2009 Feb;26(2):145-51. doi: 10.1055/s-0028-1095179. Epub 2008 Oct 31. PMID 18979408
- [Background] Lindenmayer JM, Schoenfeld S, O'Grady R, Carney JK. Methicillin-resistant Staphylococcus aureus in a high school wrestling team and the surrounding community. Arch Intern Med. 1998 Apr 27;158(8):895-9. doi: 10.1001/archinte.158.8.895. PMID 9570176
- [Background] Lindberg E, Adlerberth I, Hesselmar B, Saalman R, Strannegard IL, Aberg N, Wold AE. High rate of transfer of Staphylococcus aureus from parental skin to infant gut flora. J Clin Microbiol. 2004 Feb;42(2):530-4. doi: 10.1128/JCM.42.2.530-534.2004. PMID 14766812
- [Background] Behari P, Englund J, Alcasid G, Garcia-Houchins S, Weber SG. Transmission of methicillin-resistant Staphylococcus aureus to preterm infants through breast milk. Infect Control Hosp Epidemiol. 2004 Sep;25(9):778-80. doi: 10.1086/502476. PMID 15484804
- [Background] Huang YC, Chao AS, Chang SD, Chen YJ, Peng MT, Sung JH, Chen CJ. Association of Staphylococcus aureus colonization in parturient mothers and their babies. Pediatr Infect Dis J. 2009 Aug;28(8):742-4. doi: 10.1097/INF.0b013e31819c132a. PMID 19633520
- [Background] Mori R, Khanna R, Pledge D, Nakayama T. Meta-analysis of physiological effects of skin-to-skin contact for newborns and mothers. Pediatr Int. 2010 Apr;52(2):161-70. doi: 10.1111/j.1442-200X.2009.02909.x. Epub 2009 Jun 11. PMID 19519670
- [Background] Gregory ML, Eichenwald EC, Puopolo KM. Seven-year experience with a surveillance program to reduce methicillin-resistant Staphylococcus aureus colonization in a neonatal intensive care unit. Pediatrics. 2009 May;123(5):e790-6. doi: 10.1542/peds.2008-1526. PMID 19403471
- [Background] Harbarth S, Dharan S, Liassine N, Herrault P, Auckenthaler R, Pittet D. Randomized, placebo-controlled, double-blind trial to evaluate the efficacy of mupirocin for eradicating carriage of methicillin-resistant Staphylococcus aureus. Antimicrob Agents Chemother. 1999 Jun;43(6):1412-6. doi: 10.1128/AAC.43.6.1412. PMID 10348762
- [Derived] Lamy Filho F, de Sousa SH, Freitas IJ, Lamy ZC, Simoes VM, da Silva AA, Barbieri MA. Effect of maternal skin-to-skin contact on decolonization of Methicillin-Oxacillin-Resistant Staphylococcus in neonatal intensive care units: a randomized controlled trial. BMC Pregnancy Childbirth. 2015 Mar 19;15:63. doi: 10.1186/s12884-015-0496-1. PMID 25880822